CLINICAL TRIAL: NCT03300388
Title: Dysfunction of Adipose Tissue in Obesity, Inflammation and Aging: Mechanisms and Effects of Physical Exercise and Omega-3 Fatty Acids.
Brief Title: Obesity, Inflammation and Aging: Effects of Physical Exercise and Omega-3 Fatty Acids.
Acronym: OBELEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Centro de Estudios, Investigación y Medicina del Deporte (Other Government); Instituto de Investigación Sanitaria de Navarra (IdiSNA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OBELEX
Record Dates: First submitted 2017-08-07; First posted 2017-10-03 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Aging; Inflammation
Keywords: Insulin resistance; Exercise; Omega-3 fatty acids; Adipose tissue
MeSH Terms: conditions — Obesity; Inflammation; Insulin Resistance; Motor Activity | interventions — Docosahexaenoic Acids; Olive Oil; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): Dietary advice for a healthy diet supplemented with placebo (olive oil).
  Interventions: Dietary Supplement: Placebo (olive oil)
- Omega-3 (Experimental): Dietary advice for a healthy diet supplemented with DHA-rich dietary supplement (providing 1.650 mg/day of DHA).
  Interventions: Dietary Supplement: Omega-3 (DHA-rich dietary supplement)
- Resistance Training (Experimental): Dietary advice for a healthy diet supplemented with placebo (olive oil) and moderate resistance training program.
  Interventions: Dietary Supplement: Placebo (olive oil); Other: Resistance training
- Omega-3 + Resistance Training (Experimental): Dietary advice for a healthy diet supplemented with a DHA-rich dietary supplement (providing 1.650 mg/day of DHA) and moderate resistance training program.
  Interventions: Dietary Supplement: Omega-3 (DHA-rich dietary supplement); Other: Resistance training

INTERVENTIONS:
Dietary Supplement: Omega-3 (DHA-rich dietary supplement) — Double-blind randomized placebo-controlled intervention with DHA-rich dietary supplement with or without resistance training program for 16 weeks.
  Arms: Omega-3; Omega-3 + Resistance Training
Dietary Supplement: Placebo (olive oil) — Double-blind randomized placebo-controlled intervention with DHA-rich dietary supplement with or without resistance training program for 16 weeks.
  Arms: Control; Resistance Training
Other: Resistance training — Double-blind randomized placebo-controlled intervention with DHA-rich dietary supplement with or without resistance training program for 16 weeks.
  Arms: Omega-3 + Resistance Training; Resistance Training

SUMMARY:
Dysfunction of adipose tissue in obesity, inflammation and aging: mechanisms and effects of physical exercise and omega-3 fatty acids.

DETAILED DESCRIPTION:
Obesity is associated with the development of metabolic diseases including type 2 diabetes and immune disorders. Obesity also leads to reduced lifespan and accelerated cellular processes similar to those of aging. On the other hand, aging is accompanied by the accumulation of visceral fat and the metabolic complications associated to obesity. Both obesity and aging have been identified as chronic, low-grade inflammation disorders. The inflammation in aging has been considered as a risk factor for the development of most of age-related diseases, and therefore for morbidity and mortality in the elderly. However, the specific mechanisms leading to inflammation in aging remain largely unknown.

Resolution of inflammation is an active process which involves production of several series of specialized pro-resolving lipid mediators such lipoxins, resolvin, protectins and maresin. The hypothesis of this trial is that the chronic inflammation associated to obesity and aging could be the result of an impaired production of these specialized pro-resolutive lipid mediators, mainly in adipose tissue. On the other hand, the investigators also propose that altered transcriptional pattern might be responsible for the development of the inflammation associated with the pathophysiology of obesity and aging. Therefore the first general aim of the current project will be to characterize the mechanisms involved in the unresolved chronic inflammation that arises during obesity and aging.

Because n-3 PUFAs (polyunsaturated fatty acids) serve as substrates for the synthesis of specialized pro-resolving lipid mediators and are important transcriptional regulators, the investigators propose that dietary supplementation with n-3 PUFAs, alone or in combination with regular physical exercise could promote the resolution of local and systemic inflammation and the subsequent metabolic disorders associated to obesity and aging. A trial in overweight/obese postmenopausal women will be carried out to characterize the potential beneficial effects of regular administration of a DHA-rich dietary supplement and/or a progressive resistance training (PRT) program on weight and fat mass loss, insulin sensitivity, inflammatory markers and gene/miRNA/lipidomic/metabolomic profile in serum and/or adipose tissue. Moreover, changes in gut microbiota will be also addressed.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women
* Age between 55 and 70 years
* Body Mass Index (BMI) between 27.5 and 35 kg/m²
* Weight unchanged (± 3 kg) for the last 3 months
* Overall physical and psychological condition that the investigator believes is in accordance with the overall aim of the study

Exclusion Criteria:

* Use of regular prescription medication: specially statins, antidiabetic drugs, menopausal hormone replacement therapy
* To suffer from any chronic metabolic condition: severe dislipidemia, type 1 or 2 diabetes, hepatic (cirrhosis), renal disease, cardiovascular disease, neuromuscular disease, arthritic disease, pulmonary disease and/or other debilitating diseases
* Food allergies and/or food intolerance expected to come up during the study
* Following special diets (Atkins, vegetarian, etc.) prior three months the start of the study
* Eating disorders
* Surgically treated obesity
* Alcohol or drug abuse

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Fat mass reduction | Week 0 (baseline)
  Evaluation of body fat mass changes induced by the different interventions, analyzed by Dual X-ray Absorptiometry (DXA).
Fat mass reduction | Week 16 (end of intervention)
  Evaluation of body fat mass changes induced by the different interventions, analyzed by Dual X-ray Absorptiometry (DXA).

SECONDARY OUTCOMES:
Evolution of fat mass reduction | Week 0 (baseline)
  Evaluation of body fat mass changes induced by the different interventions analyzed by bioimpedance.
Evolution of fat mass reduction | Week 2
  Evaluation of body fat mass changes induced by the different interventions analyzed by bioimpedance.
Evolution of fat mass reduction | Week 4
  Evaluation of body fat mass changes induced by the different interventions analyzed by bioimpedance.
Evolution of fat mass reduction | Week 6
  Evaluation of body fat mass changes induced by the different interventions analyzed by bioimpedance.
Evolution of fat mass reduction | Week 8
  Evaluation of body fat mass changes induced by the different interventions analyzed by bioimpedance.
Evolution of fat mass reduction | Week 10
  Evaluation of body fat mass changes induced by the different interventions analyzed by bioimpedance.
Evolution of fat mass reduction | Week 12
  Evaluation of body fat mass changes induced by the different interventions analyzed by bioimpedance.
Evolution of fat mass reduction | Week 14
  Evaluation of body fat mass changes induced by the different interventions analyzed by bioimpedance.
Evolution of fat mass reduction | Week 16 (end of intervention)
  Evaluation of body fat mass changes induced by the different interventions analyzed by bioimpedance.
Weight loss | Week 0 (baseline)
  Changes in body weight will be measured by a body weight scale to the nearest 0.1 kg
Weight loss | Week 2
  Changes in body weight will be measured by a body weight scale to the nearest 0.1 kg
Weight loss | Week 4
  Changes in body weight will be measured by a body weight scale to the nearest 0.1 kg
Weight loss | Week 6
  Changes in body weight will be measured by a body weight scale to the nearest 0.1 kg
Weight loss | Week 8
  Changes in body weight will be measured by a body weight scale to the nearest 0.1 kg
Weight loss | Week 10
  Changes in body weight will be measured by a body weight scale to the nearest 0.1 kg
Weight loss | Week 12
  Changes in body weight will be measured by a body weight scale to the nearest 0.1 kg
Weight loss | Week 14
  Changes in body weight will be measured by a body weight scale to the nearest 0.1 kg
Weight loss | Week 16 (end of intervention)
  Changes in body weight will be measured by a body weight scale to the nearest 0.1 kg
Evolution of body composition | Week 0 (baseline)
  Evaluation of fat-free mass changes will be analyzed by bioimpedance.
Evolution of body composition | Week 2
  Evaluation of fat-free mass changes will be analyzed by bioimpedance.
Evolution of body composition | Week 4
  Evaluation of fat-free mass changes will be analyzed by bioimpedance.
Evolution of body composition | Week 6
  Evaluation of fat-free mass changes will be analyzed by bioimpedance.
Evolution of body composition | Week 8
  Evaluation of fat-free mass changes will be analyzed by bioimpedance.
Evolution of body composition | Week 10
  Evaluation of fat-free mass changes will be analyzed by bioimpedance.
Evolution of body composition | Week 12
  Evaluation of fat-free mass changes will be analyzed by bioimpedance.
Evolution of body composition | Week 14
  Evaluation of fat-free mass changes will be analyzed by bioimpedance.
Evolution of body composition | Week 16 (end of intervention)
  Evaluation of fat-free mass changes will be analyzed by bioimpedance.
Hip circumference | Week 0 (baseline)
  Hip circumference will be measured with a measuring tape.
Hip circumference | Week 8
  Hip circumference will be measured with a measuring tape.
Hip circumference | Week 16 (end of intervention)
  Hip circumference will be measured with a measuring tape.
Neck circumference | Week 0 (baseline)
  Neck circumference will be measured with a measuring tape.
Neck circumference | Week 8
  Neck circumference will be measured with a measuring tape.
Neck circumference | Week 16 (end of intervention)
  Neck circumference will be measured with a measuring tape.
Waist circumference | Week 0 (baseline)
  Waist circumference will be measured with a measuring tape.
Waist circumference | Week 8
  Waist circumference will be measured with a measuring tape.
Waist circumference | Week 16 (end of intervention)
  Waist circumference will be measured with a measuring tape.
Abdomen circumference | Week 0 (baseline)
  Abdomen circumference will be measured with a measuring tape.
Abdomen circumference | Week 8
  Abdomen circumference will be measured with a measuring tape.
Abdomen circumference | Week 16 (end of intervention)
  Abdomen circumference will be measured with a measuring tape.
Arm circumference | Week 0 (baseline)
  Arm circumference will be measured with a measuring tape.
Arm circumference | Week 8
  Arm circumference will be measured with a measuring tape.
Arm circumference | Week 16 (end of intervention)
  Arm circumference will be measured with a measuring tape.
Midthigh circumference | Week 0 (baseline)
  Midthigh circumference will be measured with a measuring tape.
Midthigh circumference | Week 8
  Midthigh circumference will be measured with a measuring tape.
Midthigh circumference | Week 16 (end of intervention)
  Midthigh circumference will be measured with a measuring tape.
Midcalf circumference | Week 0 (baseline)
  Midcalf circumference will be measured with a measuring tape.
Midcalf circumference | Week 8
  Midcalf circumference will be measured with a measuring tape.
Midcalf circumference | Week 16 (end of intervention)
  Midcalf circumference will be measured with a measuring tape.
Triceps skinfold | Week 0 (baseline)
  Triceps skinfold will be measured with a caliper.
Triceps skinfold | Week 8
  Triceps skinfold will be measured with a caliper.
Triceps skinfold | Week 16 (end of intervention)
  Triceps skinfold will be measured with a caliper.
Thigh skinfold | Week 0 (baseline)
  Thigh skinfold will be measured with a caliper.
Thigh skinfold | Week 8
  Thigh skinfold will be measured with a caliper.
Thigh skinfold | Week 16 (end of intervention)
  Thigh skinfold will be measured with a caliper.
Medial calf skinfold | Week 0 (baseline)
  Medial calf skinfold will be measured with a caliper.
Medial calf skinfold | Week 8
  Medial calf skinfold will be measured with a caliper.
Medial calf skinfold | Week 16 (end of intervention)
  Medial calf skinfold will be measured with a caliper.
Blood pressure | Week 0 (baseline)
  Systolic and diastolic blood pressure will be measured with a tensiometer.
Blood pressure | Week 8
  Systolic and diastolic blood pressure will be measured with a tensiometer.
Blood pressure | Week 16 (end of intervention)
  Systolic and diastolic blood pressure will be measured with a tensiometer.
Serum glucose | Week 0 (baseline)
  Fasting serum glucose will be measured after overnight fast.
Serum glucose | Week 16 (end of intervention)
  Fasting serum glucose will be measured after overnight fast.
Serum insulin | Week 0 (baseline)
  Fasting serum insulin will be measured after overnight fast.
Serum insulin | Week 16 (end of intervention)
  Fasting serum insulin will be measured after overnight fast.
Oral Glucose Tolerance Test | Week 0 (baseline)
  Oral Glucose Tolerance Test will be carried out after overnight fast.
Oral Glucose Tolerance Test | Week 16 (end of intervention)
  Oral Glucose Tolerance Test will be carried out after overnight fast.
Lipid metabolism biomarkers | Week 0 (baseline)
  Serum free fatty acids, triglycerides, total cholesterol, LDL-cholesterol and HDL-cholesterol concentrations will be measured after an overnight fast.
Lipid metabolism biomarkers | Week 16 (end of intervention)
  Serum free fatty acids, triglycerides, total cholesterol, LDL-cholesterol and HDL-cholesterol concentrations will be measured after an overnight fast.
Ketone bodies | Week 0 (baseline)
  Ketone bodies concentrations will be measured after an overnight fast.
Ketone bodies | Week 16 (end of intervention)
  Ketone bodies concentrations will be measured after an overnight fast.
Thyroid function (body metabolism) | Week 0 (baseline)
  TSH (thyroid-stimulating hormone), T3 and T4 hormones will be evaluated with ELISA kits
Thyroid function (body metabolism) | Week 16 (end of intervention)
  TSH (thyroid-stimulating hormone), T3 and T4 hormones will be evaluated with ELISA kits
Cardiovascular risk biomarkers | Week 0 (baseline)
  PAI-1 (plasminogen activator inhibitor-1), ADMA (asymmetric dimethylarginine) and VEGF (vascular endothelial growth factor) will be measured in plasma using ELISA kits
Cardiovascular risk biomarkers | Week 16 (end of intervention)
  PAI-1 (plasminogen activator inhibitor-1), ADMA (asymmetric dimethylarginine) and VEGF (vascular endothelial growth factor) will be measured in plasma using ELISA kits
Inflammation biomarkers | Week 0 (baseline)
  TNF-α (tumour necrosis factor-alpha), IL-6 (interleukin 6), C-reactive protein, serum A-amyloid, leptin, adiponectin, chemerin will be measured by ELISA kits
Inflammation biomarkers | Week 16 (end of intervention)
  TNF-α (tumour necrosis factor-alpha), IL-6 (interleukin 6), C-reactive protein, serum A-amyloid, leptin, adiponectin, chemerin will be measured in plasma by ELISA kits
Satiety and eating behavior traits | Week 0 (baseline)
  Satiety will be also estimated by using a VAS (visual analogue scale) questionnaire and eating behavior traits will be also evaluated with validated questionnaires
Satiety and eating behavior traits | Week 16 (end of intervention)
  Satiety will be also estimated by using a VAS (visual analogue scale) questionnaire and eating behavior traits will be also evaluated with validated questionnaires
Plasma adipokines and myo-kines | Week 0 (baseline)
  CT-1, irisin, FGF21 (fibroblast growth factor 21) and meteorin-like will be measured using ELISA kits
Plasma adipokines and myo-kines | Week 16 (end of intervention)
  CT-1, irisin, FGF21 (fibroblast growth factor 21) and meteorin-like will be measured using ELISA kits
Plasma lipids and bioactive lipid mediators | Week 0 (baseline)
  Lipidomic profile will be measured using targeted metabolomic-lipidomics by HPLC-MS (high pressure liquid chromatography-mass spectrometry).
Plasma lipids and bioactive lipid mediators | Week 16 (end of intervention)
  Lipidomic profile will be measured using targeted metabolomic-lipidomics by HPLC-MS (high pressure liquid chromatography-mass spectrometry).
Adipose tissue gene profiling | Week 0 (baseline)
  A biopsy (2 g) of subcutaneous abdominal periumbilical area adipose tissue will be obtained by liposuction under local anesthesia. RNA expression will be measured by RNA-seq or GeneChip Human Gene 2.1 ST Array (Affymetrix).
Adipose tissue gene profiling | Week 16 (end of intervention)
  A biopsy (2 g) of subcutaneous abdominal periumbilical area adipose tissue will be obtained by liposuction under local anesthesia. RNA expression will be measured by RNA-seq or GeneChip Human Gene 2.1 ST Array (Affymetrix).
Adipose tissue miRNA profiling | Week 0 (baseline)
  MiRNA expression will be measured by RNA-seq or GeneChip miRNA 4.0 Array (Affymetrix) in subcutaneous abdominal adipose tissue biopsies.
Adipose tissue miRNA profiling | Week 16 (end of intervention)
  MiRNA expression will be measured by RNA-seq or GeneChip miRNA 4.0 Array (Affymetrix) in subcutaneous abdominal adipose tissue biopsies.
Bioactive lipid mediators involved in inflammation in adipose tissue | Week 0 (baseline)
  Lipidomic profile will be measured using targeted metabolomic-lipidomics by HPLC-MS
Bioactive lipid mediators involved in inflammation in adipose tissue | Week 16 (end of intervention)
  Lipidomic profile will be measured using targeted metabolomic-lipidomics by HPLC-MS
Determination of telomeres length | Week 0 (baseline)
  Telomeres length will be measured in genomic DNA extracted from human peripheral blood and adipose tissue samples with a real-time quantitative PCR (polymerase chain reaction) approach.
Determination of telomeres length | Week 16 (end of intervention)
  Telomeres length will be measured in genomic DNA extracted from human peripheral blood and adipose tissue samples with a real-time quantitative PCR (polymerase chain reaction) approach.
Characterization of gut microbiota | Week 0 (baseline)
  Feces will collected and gut microbiota profiling will be carried out by high-throughput 16S (Svedberg units) rDNA (ribosomal deoxyribonucleic acid) amplicon sequencing approach.
Characterization of gut microbiota | Week 16 (end of intervention)
  Feces will collected and gut microbiota profiling will be carried out by high-throughput 16S (Svedberg units) rDNA (ribosomal deoxyribonucleic acid) amplicon sequencing approach.
Urine metabolomic profile | Week 0 (baseline)
  Urine will be collected and urinary metabolomic profile will be also evaluated by a HPLC-MS approach.
Urine metabolomic profile | Week 16 (end of intervention)
  Urine will be collected and urinary metabolomic profile will be also evaluated by a HPLC-MS approach.

CONTACTS AND LOCATIONS:
Overall Officials: María J Moreno-Aliaga, PhD, Principal Investigator — University of Navarra; Silvia Lorente-Cebrián, PhD, Principal Investigator — University of Navarra
Locations (1):
- Department of Nutrition, Food Science and Physiology. Centre for Nutrition Research., Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Fernandez L, Gonzalez-Muniesa P, Laiglesia LM, Sainz N, Prieto-Hontoria PL, Escote X, Odriozola L, Corrales FJ, Arbones-Mainar JM, Martinez JA, Moreno-Aliaga MJ. Maresin 1 improves insulin sensitivity and attenuates adipose tissue inflammation in ob/ob and diet-induced obese mice. FASEB J. 2017 May;31(5):2135-2145. doi: 10.1096/fj.201600859R. Epub 2017 Feb 10. PMID 28188173
- [Background] Lopez-Yoldi M, Stanhope KL, Garaulet M, Chen XG, Marcos-Gomez B, Carrasco-Benso MP, Santa Maria EM, Escote X, Lee V, Nunez MV, Medici V, Martinez-Anso E, Sainz N, Huerta AE, Laiglesia LM, Prieto J, Martinez JA, Bustos M, Havel PJ, Moreno-Aliaga MJ. Role of cardiotrophin-1 in the regulation of metabolic circadian rhythms and adipose core clock genes in mice and characterization of 24-h circulating CT-1 profiles in normal-weight and overweight/obese subjects. FASEB J. 2017 Apr;31(4):1639-1649. doi: 10.1096/fj.201600396RR. Epub 2017 Jan 17. PMID 28096235
- [Background] Laiglesia LM, Lorente-Cebrian S, Prieto-Hontoria PL, Fernandez-Galilea M, Ribeiro SM, Sainz N, Martinez JA, Moreno-Aliaga MJ. Eicosapentaenoic acid promotes mitochondrial biogenesis and beige-like features in subcutaneous adipocytes from overweight subjects. J Nutr Biochem. 2016 Nov;37:76-82. doi: 10.1016/j.jnutbio.2016.07.019. Epub 2016 Aug 26. PMID 27637001
- [Background] Huerta AE, Prieto-Hontoria PL, Fernandez-Galilea M, Escote X, Martinez JA, Moreno-Aliaga MJ. Effects of dietary supplementation with EPA and/or alpha-lipoic acid on adipose tissue transcriptomic profile of healthy overweight/obese women following a hypocaloric diet. Biofactors. 2017 Jan 2;43(1):117-131. doi: 10.1002/biof.1317. Epub 2016 Aug 10. PMID 27507611
- [Background] Huerta AE, Prieto-Hontoria PL, Sainz N, Martinez JA, Moreno-Aliaga MJ. Supplementation with alpha-Lipoic Acid Alone or in Combination with Eicosapentaenoic Acid Modulates the Inflammatory Status of Healthy Overweight or Obese Women Consuming an Energy-Restricted Diet. J Nutr. 2015 Apr 1;146(4):889S-896S. doi: 10.3945/jn.115.224105. PMID 26962183
- [Background] Milagro FI, Moreno-Aliaga MJ, Martinez JA. FTO Obesity Variant and Adipocyte Browning in Humans. N Engl J Med. 2016 Jan 14;374(2):190-1. doi: 10.1056/NEJMc1513316. No abstract available. PMID 26760097
- [Background] Prieto-Hontoria PL, Perez-Matute P, Fernandez-Galilea M, Lopez-Yoldi M, Sinal CJ, Martinez JA, Moreno-Aliaga MJ. Effects of alpha-lipoic acid on chemerin secretion in 3T3-L1 and human adipocytes. Biochim Biophys Acta. 2016 Mar;1861(3):260-8. doi: 10.1016/j.bbalip.2015.12.011. Epub 2015 Dec 22. PMID 26721419
- [Background] Martinez-Fernandez L, Laiglesia LM, Huerta AE, Martinez JA, Moreno-Aliaga MJ. Omega-3 fatty acids and adipose tissue function in obesity and metabolic syndrome. Prostaglandins Other Lipid Mediat. 2015 Sep;121(Pt A):24-41. doi: 10.1016/j.prostaglandins.2015.07.003. Epub 2015 Jul 26. PMID 26219838
- [Background] Mansego ML, Milagro FI, Zulet MA, Moreno-Aliaga MJ, Martinez JA. Differential DNA Methylation in Relation to Age and Health Risks of Obesity. Int J Mol Sci. 2015 Jul 24;16(8):16816-32. doi: 10.3390/ijms160816816. PMID 26213922
- [Background] Huerta AE, Prieto-Hontoria PL, Fernandez-Galilea M, Sainz N, Cuervo M, Martinez JA, Moreno-Aliaga MJ. Circulating irisin and glucose metabolism in overweight/obese women: effects of alpha-lipoic acid and eicosapentaenoic acid. J Physiol Biochem. 2015 Sep;71(3):547-58. doi: 10.1007/s13105-015-0400-5. Epub 2015 Mar 28. PMID 25820474
- [Background] Lorente-Cebrian S, Costa AG, Navas-Carretero S, Zabala M, Laiglesia LM, Martinez JA, Moreno-Aliaga MJ. An update on the role of omega-3 fatty acids on inflammatory and degenerative diseases. J Physiol Biochem. 2015 Jun;71(2):341-9. doi: 10.1007/s13105-015-0395-y. Epub 2015 Mar 11. PMID 25752887
- [Background] Huerta AE, Navas-Carretero S, Prieto-Hontoria PL, Martinez JA, Moreno-Aliaga MJ. Effects of alpha-lipoic acid and eicosapentaenoic acid in overweight and obese women during weight loss. Obesity (Silver Spring). 2015 Feb;23(2):313-21. doi: 10.1002/oby.20966. Epub 2014 Dec 31. PMID 25594166
- [Background] Gonzalez-Muniesa P, Marrades MP, Martinez JA, Moreno-Aliaga MJ. Differential proinflammatory and oxidative stress response and vulnerability to metabolic syndrome in habitual high-fat young male consumers putatively predisposed by their genetic background. Int J Mol Sci. 2013 Aug 22;14(9):17238-55. doi: 10.3390/ijms140917238. PMID 23975165
- [Background] Lorente-Cebrian S, Costa AG, Navas-Carretero S, Zabala M, Martinez JA, Moreno-Aliaga MJ. Role of omega-3 fatty acids in obesity, metabolic syndrome, and cardiovascular diseases: a review of the evidence. J Physiol Biochem. 2013 Sep;69(3):633-51. doi: 10.1007/s13105-013-0265-4. Epub 2013 Jun 22. PMID 23794360
- [Background] Lorente-Cebrian S, Bustos M, Marti A, Fernandez-Galilea M, Martinez JA, Moreno-Aliaga MJ. Eicosapentaenoic acid inhibits tumour necrosis factor-alpha-induced lipolysis in murine cultured adipocytes. J Nutr Biochem. 2012 Mar;23(3):218-27. doi: 10.1016/j.jnutbio.2010.11.018. Epub 2011 Apr 14. PMID 21497077
- [Background] Marrades MP, Gonzalez-Muniesa P, Martinez JA, Moreno-Aliaga MJ. A dysregulation in CES1, APOE and other lipid metabolism-related genes is associated to cardiovascular risk factors linked to obesity. Obes Facts. 2010 Oct;3(5):312-8. doi: 10.1159/000321451. Epub 2010 Oct 15. PMID 20975297
- [Background] Marrades MP, Gonzalez-Muniesa P, Arteta D, Martinez JA, Moreno-Aliaga MJ. Orchestrated downregulation of genes involved in oxidative metabolic pathways in obese vs. lean high-fat young male consumers. J Physiol Biochem. 2011 Mar;67(1):15-26. doi: 10.1007/s13105-010-0044-4. Epub 2010 Sep 30. PMID 20882379
- [Background] Moreno-Aliaga MJ, Lorente-Cebrian S, Martinez JA. Regulation of adipokine secretion by n-3 fatty acids. Proc Nutr Soc. 2010 Aug;69(3):324-32. doi: 10.1017/S0029665110001801. Epub 2010 Jun 14. PMID 20540825
- [Background] Lorente-Cebrian S, Bustos M, Marti A, Martinez JA, Moreno-Aliaga MJ. Eicosapentaenoic acid up-regulates apelin secretion and gene expression in 3T3-L1 adipocytes. Mol Nutr Food Res. 2010 May;54 Suppl 1:S104-11. doi: 10.1002/mnfr.200900522. PMID 20352620
- [Background] Lorente-Cebrian S, Bustos M, Marti A, Martinez JA, Moreno-Aliaga MJ. Eicosapentaenoic acid stimulates AMP-activated protein kinase and increases visfatin secretion in cultured murine adipocytes. Clin Sci (Lond). 2009 Aug 14;117(6):243-9. doi: 10.1042/CS20090020. PMID 19296827
- [Background] Perez-Echarri N, Perez-Matute P, Marcos-Gomez B, Marti A, Martinez JA, Moreno-Aliaga MJ. Down-regulation in muscle and liver lipogenic genes: EPA ethyl ester treatment in lean and overweight (high-fat-fed) rats. J Nutr Biochem. 2009 Sep;20(9):705-14. doi: 10.1016/j.jnutbio.2008.06.013. Epub 2008 Sep 30. PMID 18829285
- See also: Centre for Nutrition Research. University of Navarra — http://www.unav.edu/web/centro-de-investigacion-en-nutricion
- See also: Department of Nutrition, Food Science and Physiology. University of Navarra — http://www.unav.edu/departamento/caft/